CLINICAL TRIAL: NCT06080984
Title: The Application of Novel Oncolytic Virus in Late Stage Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Professor, West China Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-833
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Malignant Tumor
Keywords: Solid Tumors; Oncolytic Virus
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Cohort 1 (Experimental): This arm includes 6 head and neck squamous cell carcinoma patients. Patients in the study receive intratumoral treatment with a novel oncolytic virus SDJ001 at two dose levels: 5x10^11 and 1x10^12 pfu per person. At the current dose levels, intratumoral injection is administered on the first day of each treatment cycle. Each treatment cycle consists of three weeks, continuing until tumor growth is observed following injection or until the patient experiences intolerable toxic effects.
  Ultrasound-guided injection may be used when necessary (2.0 mL for tumors with a diameter >2.5 cm, 1.0 mL for diameters of 1.5-2.5 cm, 0.5 mL for diameters of 0.5-1.5 cm, and 0.1 mL for diameters <0.5 cm, with a maximum of 4 mL).
  Interventions: Drug: Oncolytic Virus SDJ001
- Treatment Cohort 2 (Experimental): This arm includes 9 melanoma patients. Patients in the study receive intratumoral treatment with a novel oncolytic virus YD06-1 at a concentration of 10^6 pfu/mL to 10^8 pfu/ml following a dose escalation plan. Each subject receives only one injection at the corresponding concentration, with the dose determined based on the size of the tumor mass. (Diameter ≤1.5 cm, maximum of 1 mL; diameter 1.5-2.5 cm, maximum of 2 mL; diameter greater than 2.5 cm, maximum of 4 mL). The second dose is administered three weeks after the first dose, followed by subsequent doses at two-week intervals.
  Interventions: Drug: Oncolytic Virus YD06-1
- Treatment Cohort 3 (Experimental): This arm includes 9 sarcoma patients. Patients in the study receive intratumoral treatment with a novel oncolytic virus YD06-1 at a concentration of 10^6 pfu/mL to 10^8 pfu/ml following a dose escalation plan. Each subject receives only one injection at the corresponding concentration, with the dose determined based on the size of the tumor mass. (Diameter ≤1.5 cm, maximum of 1 mL; diameter 1.5-2.5 cm, maximum of 2 mL; diameter greater than 2.5 cm, maximum of 4 mL). The second dose is administered three weeks after the first dose, followed by subsequent doses at two-week intervals.
  Interventions: Drug: Oncolytic Virus YD06-1

INTERVENTIONS:
Drug: Oncolytic Virus SDJ001 — Patients in the study receive intratumoral treatment with SDJ001 at two dose levels: 5x10^11 and 1x10^12 pfu per person. At the current dose levels, intratumoral injection is administered on the first day of each treatment cycle. Each treatment cycle consists of three weeks, continuing until tumor growth is observed following injection or until the patient experiences intolerable toxic effects.
  Ultrasound-guided injection may be used when necessary (2.0 mL for tumors with a diameter >2.5 cm, 1.0 mL for diameters of 1.5-2.5 cm, 0.5 mL for diameters of 0.5-1.5 cm, and 0.1 mL for diameters <0.5 cm, with a maximum of 4 mL).
  Arms: Treatment Cohort 1
Drug: Oncolytic Virus YD06-1 — Patients in the study receive intratumoral treatment with a novel oncolytic virus YD06-1 at a concentration of 10^6 pfu/mL to 10^8 pfu/ml following a dose escalation plan. Each subject receives only one injection at the corresponding concentration, with the dose determined based on the size of the tumor mass. (Diameter ≤1.5 cm, maximum of 1 mL; diameter 1.5-2.5 cm, maximum of 2 mL; diameter greater than 2.5 cm, maximum of 4 mL). The second dose is administered three weeks after the first dose, followed by subsequent doses at two-week intervals.
  Arms: Treatment Cohort 2; Treatment Cohort 3

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of novel oncolytic virus in late stage solid tumors.

DETAILED DESCRIPTION:
Oncolytic viruses (OVs) are naturally occurring or recombinant viruses that can selectively destroy tumor cells without harming normal cells. After infecting the host, oncolytic viruses can replicate within host cells, and the progeny viruses released can further infect neighboring host cells and kill the tumor while triggering local or systemic anti-tumor immune responses. Compared to traditional treatments, oncolytic virus therapy offers advantages such as good targeting, minimal adverse reactions, multiple tumor-killing pathways, and reduced likelihood of developing resistance.

Several clinical studies have found that oncolytic viruses can provide clinical benefits to patients with different types, stages, and even advanced metastatic tumors. Importantly, when used in combination with radiation therapy or chemotherapy, they exhibit good synergistic effects. Especially when used in combination with immunotherapy, oncolytic viruses can sensitize tumor types that were initially unresponsive to immune checkpoint inhibitors.

Currently, oncolytic viruses are believed to exert anti-tumor activity through three main mechanisms:

1. Direct Oncolytic Effect:

   Oncolytic viruses can undergo specific replication within tumor cells, primarily due to the tumor's specific genetic alterations that prevent the cell's signaling pathways from sensing and blocking virus replication. Tumor interferon defects prevent the regulation of the virus defense system, increasing sensitivity to virus infection. By genetic modification, the virulence factors of oncolytic viruses can be weakened or deleted, preventing virus replication in normal tissues while retaining the ability to replicate within tumor cells and kill them.
2. Elicitation of Anti-Tumor Immune Responses:

   Oncolytic virus infection of tumor cells can transform "cold" tumors into "hot" tumors, thereby triggering local and systemic anti-tumor immune responses. Immune suppressive factors in the tumor microenvironment, such as regulatory lymphocytes, interleukin-10 (IL-10), and programmed death-ligand 1 (PD-L1), can protect tumors from immune surveillance. Oncolytic viruses disrupt the existing tissue structure in the tumor microenvironment and can reverse the immunosuppressive microenvironment, transitioning it from immune suppression to immune activation. After oncolytic virus infection of tumor cells, cell lysis occurs, releasing tumor-associated antigens, activating dendritic cells, increasing the infiltration of cytotoxic T lymphocytes, and recruiting other immune-related cells and molecules. This results in an increase in tumor-specific immune responses, leading to the clearance of distant and uninfected tumor cells.
3. Expression of Anti-Tumor Target Genes and Anti-Angiogenesis:

Through genetic engineering, oncolytic viruses can express target genes that have anti-tumor effects, such as P53, GM-CSF, IL-12, IL-15, anti-PD-L1, etc., further enhancing their anti-tumor effects. In addition, some oncolytic viruses can infect and destroy the tumor's vascular system, inducing neutrophil infiltration, leading to vascular collapse and tumor cell death.

Oncolytic viruses (OVs) can be categorized into DNA virus carriers and RNA virus carriers based on the type of nucleic acid in their genomes. DNA viruses mainly include herpes simplex virus (HSV), adenovirus (AdV), vaccinia virus (VV), and parvovirus H1; while RNA viruses mainly include reovirus (RV), Coxsackievirus (CV), poliovirus (PV), measles virus (MV), Newcastle disease virus (NDV), and vesicular stomatitis virus (VSV). Among them, the five most commonly used oncolytic viruses in clinical research are adenovirus, HSV-1, reovirus, vaccinia virus, and Newcastle disease virus.

To date, five oncolytic virus products have been approved for marketing globally. There are hundreds of projects in clinical trial stages, especially in recent years, new generations of oncolytic viruses developed and marketed or in clinical stages have shown better safety and stronger anti-tumor capabilities.

Our project team has isolated and modified multiple strains of genetically engineered oncolytic herpes viruses, selecting the best strains for in vivo and in vitro pharmacological and safety evaluations. We have achieved anti-tumor effects superior to currently approved oncolytic virus control drugs. This virus has been engineered to delete virulence factors that are toxic to normal cells, and genetic engineering modifications have been made at multiple genomic loci. It can selectively replicate in tumor cells and can express recombinant bispecific antibodies at high levels. Compared to existing oncolytic virus formulations, this virus demonstrates improved safety and anti-tumor activity and holds great promise for clinical translation. In preliminary studies, the project team has also demonstrated significant anti-tumor effects of oncolytic adenovirus expressing this bispecific antibody. Therefore, in this clinical trial, our project team plans to conduct clinical translational research using the original strain based on proprietary intellectual property that has undergone genetic engineering improvements.

The implementation of this project will provide a highly potential and hopeful clinical treatment strategy for advanced cancer patients with no other treatment options. It will also provide new ideas, strategies, and experimental evidence for the development of oncolytic virus new drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: ≥18 years.
2. a)Patients with confirmed advanced squamous cell carcinoma of the head and neck (including nasopharynx) who meet the following criteria: Patients who have failed standard second-line treatment. Tumors that cannot be cured through local treatment (surgery or definitive radiation therapy).

   b)Patients with stage III malignant melanoma who are not eligible for surgical resection, or patients with stage IV malignant melanoma, who have failed at least two lines of standard treatment (including chemotherapy, immunotherapy or targeted therapy).

   c)Patients with locally unresectable or metastatic advanced soft tissue sarcomas, who have failed prior systemic treatments.
3. ECOG performance status score: 0-1.
4. Expected survival ≥3 months.
5. Time since the last chemotherapy/radiotherapy/surgery is more than 28 days.
6. Adequate organ function, as defined by the following criteria within 14 days before enrollment:

   Hematology: Hemoglobin ≥90g/L (without blood transfusion in the last 14 days); Neutrophil count >1.5×10^9/L; Platelet count ≥80×10^9/L.

   Biochemistry: Total bilirubin ≤1.5×ULN (upper limit of normal); Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤2.5×ULN; if there is liver metastasis, ALT or AST ≤5×ULN; Estimated glomerular filtration rate ≥60ml/min (Cockcroft-Gault formula).

   Cardiac Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%.
7. Patients with injectable lesions (those suitable for direct injection or injection with the assistance of medical imaging), defined as follows: at least one injectable lesion in the skin, mucous membrane, subcutaneous tissue, or lymph node with a longest diameter ≥10 mm, or multiple injectable lesions with a total longest diameter ≥10 mm
8. No continuing acute toxic effects of any prior radiotherapy, chemotherapy, or surgical intervention, i.e., all such effects must have resolved to Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0) Grade 1.
9. Signed written informed consent Subjects must sign a written informed consent form approved by the competent authority and the research institution and date it. The informed consent form must be signed before any protocol-related procedures (not part of the subject's routine medical care) are conducted.

Subjects must be willing and able to comply with the scheduled visits, treatment regimen, laboratory tests, and other requirements of the study.

Exclusion Criteria:

1. Participated in another drug clinical trial within the past 4 weeks.
2. Tumor located near major blood vessels or the trachea.
3. Has poorly controlled clinical heart symptoms or diseases, such as NYHA class 2 or higher heart failure, unstable angina, myocardial infarction within the past year, clinically significant ventricular or supraventricular arrhythmias requiring treatment or intervention.
4. For female subjects: pregnant or lactating women.
5. Persistent or active infections, including but not limited to: active pulmonary tuberculosis, positive HIV (Human Immunodeficiency Virus) antibodies, positive HBsAg (Hepatitis B Surface Antigen), positive HBcAb (Hepatitis B Core Antibody), and positive HCV (Hepatitis C Virus) antibody test results.

   1. Participants who are positive for HBsAg and/or HBcAb must also provide baseline HBV DNA results and undergo HBV DNA monitoring during the treatment according to the protocol.
   2. Participants with HBV DNA results of 10^4 copies/ml or ≥ 2000 IU/mL and any of the following conditions should be excluded: 1) positive results for HBsAg and/or HBeAg; 2) positive results for HBcAb and negative results for all others.
   3. Patients with a positive HCV antibody test result are only ineligible for study participation if their HCV RNA test result is positive..
6. Has a history of substance abuse that cannot be discontinued or has psychiatric disorders.
7. Has any active autoimmune disease or a history of autoimmune disease, including but not limited to uveitis, enteritis, pituitary inflammation, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or childhood asthma that has completely resolved in adulthood without the need for intervention may be included; subjects with asthma requiring bronchodilators for medical intervention cannot be included.
8. Patients who have used systemic corticosteroids (>10g/day of prednisone or an equivalent dose) or other immunosuppressive drugs in the 4 weeks prior to the initial administration of the study drug will be excluded.
9. Has a history of substance abuse or known medical, psychological, or social conditions, such as a history of alcoholism or drug abuse.
10. Known allergy, hypersensitivity reaction, or intolerance to oncolytic virus research (including any excipients). A history of severe allergies to any drugs, foods, or vaccines, such as anaphylactic shock, angioedema, respiratory distress, purpura, thrombocytopenic purpura, or localized allergic necrotizing reaction (Arthus reaction), etc.
11. Female subjects with pregnancy plans during the screening period or male subjects with partners who have pregnancy plans.
12. Has accompanying diseases judged by the investigator to be seriously harmful to patient safety or affecting the patient's completion of the study.
13. Patients who have undergone major surgery other than diagnosis or have unhealed wounds, ulcers, or fractures within the 28 days prior to the initial administration of the investigational drug will be excluded. For patients with lesion rupture, screening may be considered, and the eligibility will be jointly assessed by the investigator and the sponsor, depending on the specific circumstances of the rupture. The injection site should be as far away from the rupture site as possible, and during the treatment period, rupture-related adverse events should not be recorded as investigational drug-related adverse events.
14. During the course of the study, the use of drugs against HSV, including but not limited to acyclovir, valacyclovir, penciclovir, famciclovir, ganciclovir, foscarnet, and cidofovir, may be required.
15. Patients with episodes of oral herpes (cold sores) may present with small, bead-like, tense vesicles on or around the lips during the initial outbreak, typically measuring approximately 0.5 to 1.5 centimeters in size. These vesicles may also appear in the nose, ear, or finger areas and are often associated with significant pain. Recurrent oral herpes typically presents as ulcers above the vermilion border of the lip (lip herpes) and occasionally as ulcers above the hard palate mucosa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 12 months
  Adverse events defined as the number of participants with adverse events

SECONDARY OUTCOMES:
Objective response rate | up to 12 months
  ORR is defined as the percentage of patients who achieve a response, which can either be complete response (complete disappearance of lesions) or partial response (reduction in the sum of maximal tumor diameters by at least 30% or more)
Progress-Free Survival | up to 12 months
  PFS is defined as the time from the administration of the first dose to first disease
Overall Survival | up to 12 months
  OS is defined as the time from the administration of the first dose to death.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Ibarra AMC, Cecatto RB, Motta LJ, Dos Santos Franco AL, de Fatima Teixeira da Silva D, Nunes FD, Hamblin MR, Rodrigues MFSD. Photodynamic therapy for squamous cell carcinoma of the head and neck: narrative review focusing on photosensitizers. Lasers Med Sci. 2022 Apr;37(3):1441-1470. doi: 10.1007/s10103-021-03462-3. Epub 2021 Dec 2. PMID 34855034
- [Background] Andtbacka RH, Kaufman HL, Collichio F, Amatruda T, Senzer N, Chesney J, Delman KA, Spitler LE, Puzanov I, Agarwala SS, Milhem M, Cranmer L, Curti B, Lewis K, Ross M, Guthrie T, Linette GP, Daniels GA, Harrington K, Middleton MR, Miller WH Jr, Zager JS, Ye Y, Yao B, Li A, Doleman S, VanderWalde A, Gansert J, Coffin RS. Talimogene Laherparepvec Improves Durable Response Rate in Patients With Advanced Melanoma. J Clin Oncol. 2015 Sep 1;33(25):2780-8. doi: 10.1200/JCO.2014.58.3377. Epub 2015 May 26. PMID 26014293
- [Background] Chesney JA, Ribas A, Long GV, Kirkwood JM, Dummer R, Puzanov I, Hoeller C, Gajewski TF, Gutzmer R, Rutkowski P, Demidov L, Arenberger P, Shin SJ, Ferrucci PF, Haydon A, Hyngstrom J, van Thienen JV, Haferkamp S, Guilera JM, Rapoport BL, VanderWalde A, Diede SJ, Anderson JR, Treichel S, Chan EL, Bhatta S, Gansert J, Hodi FS, Gogas H. Randomized, Double-Blind, Placebo-Controlled, Global Phase III Trial of Talimogene Laherparepvec Combined With Pembrolizumab for Advanced Melanoma. J Clin Oncol. 2023 Jan 20;41(3):528-540. doi: 10.1200/JCO.22.00343. Epub 2022 Aug 23. PMID 35998300
- [Background] Harrington KJ, Kong A, Mach N, Chesney JA, Fernandez BC, Rischin D, Cohen EEW, Radcliffe HS, Gumuscu B, Cheng J, Snyder W, Siu LL. Talimogene Laherparepvec and Pembrolizumab in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (MASTERKEY-232): A Multicenter, Phase 1b Study. Clin Cancer Res. 2020 Oct 1;26(19):5153-5161. doi: 10.1158/1078-0432.CCR-20-1170. Epub 2020 Jul 15. PMID 32669371
- [Background] Twumasi-Boateng K, Pettigrew JL, Kwok YYE, Bell JC, Nelson BH. Oncolytic viruses as engineering platforms for combination immunotherapy. Nat Rev Cancer. 2018 Jul;18(7):419-432. doi: 10.1038/s41568-018-0009-4. PMID 29695749
- [Background] Xia ZJ, Chang JH, Zhang L, Jiang WQ, Guan ZZ, Liu JW, Zhang Y, Hu XH, Wu GH, Wang HQ, Chen ZC, Chen JC, Zhou QH, Lu JW, Fan QX, Huang JJ, Zheng X. [Phase III randomized clinical trial of intratumoral injection of E1B gene-deleted adenovirus (H101) combined with cisplatin-based chemotherapy in treating squamous cell cancer of head and neck or esophagus]. Ai Zheng. 2004 Dec;23(12):1666-70. Chinese. PMID 15601557
- [Background] Ribas A, Dummer R, Puzanov I, VanderWalde A, Andtbacka RHI, Michielin O, Olszanski AJ, Malvehy J, Cebon J, Fernandez E, Kirkwood JM, Gajewski TF, Chen L, Gorski KS, Anderson AA, Diede SJ, Lassman ME, Gansert J, Hodi FS, Long GV. Oncolytic Virotherapy Promotes Intratumoral T Cell Infiltration and Improves Anti-PD-1 Immunotherapy. Cell. 2018 Aug 9;174(4):1031-1032. doi: 10.1016/j.cell.2018.07.035. No abstract available. PMID 30096300
- [Background] Goradel NH, Baker AT, Arashkia A, Ebrahimi N, Ghorghanlu S, Negahdari B. Oncolytic virotherapy: Challenges and solutions. Curr Probl Cancer. 2021 Feb;45(1):100639. doi: 10.1016/j.currproblcancer.2020.100639. Epub 2020 Aug 15. PMID 32828575